CLINICAL TRIAL: NCT04798885
Title: Interdisciplinary Intervention for Patients With Post-concussion Symptoms 3-6 Months Post-injury (GAIN 2.0). A Stepped Wedge Cluster Randomised Trial: Effect on Symptoms, Participation in Daily Activities, and Labour Market Attachment
Brief Title: Get Going After concussioN 2.0
Acronym: GAIN2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Sygeforsikringen danmark (Unknown); Hammel Neurorehabilitation Centre and University Research Clinic (Other); Municipalities in Central Denmark Region (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAIN 2.0
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Commotio Cerebri; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (No Intervention): Participants will be informed about typical Post Concussion Symptoms and the process of typical recovery as well as given reassurance concerning the prognosis. Advice concerning the use of pain relief medication will also be provided.
- GAIN 2.0 intervention (Experimental): An eight-week, interdisciplinary intervention program based on principles from cognitive behavioural therapy (CBT) and gradual return to activities.
  Interventions: Behavioral: GAIN 2.0

INTERVENTIONS:
Behavioral: GAIN 2.0 — 1) three structured group sessions of two hours duration performed jointly by a neuropsychologist, an occupational therapist and a physiotherapist. Relatives are also invited. 2) Up to five weekly semi-structured individual sessions of 30 min. duration with an allocated therapist
  Arms: GAIN 2.0 intervention

SUMMARY:
The study tests the promising results of a previous study (GAIN 1.0) in a larger RCT (GAIN 2.0) which takes place in the municipalities of Central Denmark Region where citizens live their daily lives and whose health- and social care systems support citizens who experience persisting PCS.

DETAILED DESCRIPTION:
Concussion, the mildest form of traumatic brain injury, is an important public health concern. Recent studies estimate that persistent post-concussion symptoms (PCS) are present in almost half of the affected citizens at one year post-injury. Prospective studies have demonstrated that these citizens are at risk of developing long-lasting symptoms which are associated with high societal burden due to long-term impact on labour market attachment and increased use of health care and social benefits. In Denmark, there has in recent years been an increasing awareness on societal impact and personal consequences of PCS. Accordingly, clinicians as well as social workers and therapists in the municipalities point to the gab in knowledge concerning PCS and advocate urgently for evidence-based treatment for these citizens. Recently, the research group behind this application developed a novel early intervention - "Get going After concussIoN" (GAIN 1.0) - for citizens who experience persistent PCS three to six months post-concussion. The intervention was tested in a randomized controlled trial (RCT) with promising results. However, it was delivered in a single hospital setting in which these citizens are normally not cared for. In this study the intention is to test the results of GAIN 1.0 in a larger RCT (GAIN 2.0) which takes place in the municipalities of Central Denmark Region where citizens live their daily lives and whose health- and social care systems support citizens who experience persisting PCS.

ELIGIBILITY:
Inclusion Criteria:

1. Concussion caused by a head trauma according to the diagnostic criteria recommended by WHO. Participants must be referred to the project within two to four months of injury.
2. Age 18 to 60 years at the time of the trauma
3. A RPQ score ≥20.
4. Able to understand, speak and read Danish.
5. Living in Central Denmark Region.

Exclusion Criteria:

1. Objective neurological findings and/or acute trauma CT scan indicating neurological disease or brain damage.
2. Previous concussion leading to persistent PCS within the last two years.
3. Severe misuse of alcohol, prescription drugs and/or illegal drugs.
4. Psychiatric morbidity or severe neurological disease that impedes participation in the program, i.e. Bipolar Disorder, autism, psychotic disorder (life time), multiple sclerosis etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of at least seven in the sum score on the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) | Three months after end of treatment
  RPQ is a self-report scale to measure the severity of Post Concussion Symptoms covering physical, cognitive, and emotional symptoms with 16 sub-items and a total sum score (range 0-64, higher score define more severe status)

SECONDARY OUTCOMES:
Sumscore in the dimension 'time spend on daily activities' on the Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P). | Three months after end of treatment
  Utrecht Scale for Evaluation of Rehabilitation-Participation is a generic measurement that both objectively and subjectively measure participation in Instrumental Activities of Daily Living (IADL) such as work, voluntary work, education, family duties and responsibilities, leisure activities, transportation, communication and social activities in three dimensions. The sumscore in each dimension is converted to a 0-100 metric with higher scores meaning af better outcome.
Sumscore in the dimension 'limitations' on the Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P) | Three months after end of treatment
  Utrecht Scale for Evaluation of Rehabilitation-Participation is a generic measurement that both objectively and subjectively measure participation in Instrumental Activities of Daily Living (IADL) such as work, voluntary work, education, family duties and responsibilities, leisure activities, transportation, communication and social activities in three dimensions.The sumscore in each dimension is converted to a 0-100 metric with higher scores meaning af better outcome.
Sumscore in the dimension 'satisfaction with participation' on the Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P) | Three months after end of treatment
  Utrecht Scale for Evaluation of Rehabilitation-Participation is a generic measurement that both objectively and subjectively measure participation in Instrumental Activities of Daily Living (IADL) such as work, voluntary work, education, family duties and responsibilities, leisure activities, transportation, communication and social activities in three dimensions.The sumscore in each dimension is converted to a 0-100 metric with higher scores meaning af better outcome.
Long term sick leave defined as public assistance benefits related to illness in more than three consecutive weeks | Within 12 months after concussion
  Calculated based on weekly public assistance benefits extracted from the DREAM register
Cumulated incidence proportion of participants on long term sick leave defined as receiving public assistance benefits related to illness in more than three consecutive weeks | Within 36 months after concussion
  Calculated based on weekly public assistance benefits extracted from the DREAM register
Proportion of employed participants defined as receiving no public assistance benefits except from state education fund grants | At 12 months after concussion
  Calculated based on weekly public assistance benefits extracted from the DREAM register
Proportion of employed participants defined as receiving no public assistance benefits except from state education fund grants | At 36 months after concussion
  Calculated based on weekly public assistance benefits extracted from the DREAM register
Degree of job stability based on whether labor market contributions have been paid | At 12 months after concussion
  Monthly measure extracted from the DREAM register
Degree of job stability based on whether labor market contributions have been paid | At 36 months after concussion
  Monthly measure extracted from the DREAM register

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Professor, Principal Investigator — Hammel Neurorehabilitation Centre and University clinic
Locations (1):
- Regionshospitalet Hammel Neurocenter, Hammel, Denmark

REFERENCES:
- [Derived] Naess-Schmidt ET, Thastum MM, Stabel HH, Odgaard L, Pedersen AR, Rask CU, Silverberg ND, Schroder A, Nielsen JF. Interdisciplinary intervention (GAIN) for adults with post-concussion symptoms: a study protocol for a stepped-wedge cluster randomised trial. Trials. 2022 Jul 29;23(1):613. doi: 10.1186/s13063-022-06572-7. PMID 35906645